CLINICAL TRIAL: NCT07030270
Title: A Clinical Trial Comparing Surfactant Administration Through Supraglottic Airway or Thin Catheter for Preterm Infants
Brief Title: Comparing Surfactant Administration Through Supraglottic Airway and Thin Catheter for Preterm Infants
Acronym: SALTI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Melody Chiu, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU20250018
Record Dates: First submitted 2025-05-29; First posted 2025-06-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Distress Syndrome (RDS); Surfactant
Keywords: preterm infants; surfactant therapy; respiratory outcomes
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surfactant Administration through Laryngeal or Supraglottic Airway (Experimental)
  Interventions: Procedure: Surfactant Administration through Laryngeal or Supraglottic Airway
- Surfactant Administration through Thin Catheter (Active Comparator)
  Interventions: Procedure: Surfactant Administration through Thin Catheter

INTERVENTIONS:
Procedure: Surfactant Administration through Laryngeal or Supraglottic Airway — Surfactant Administration through Supraglottic Airway Devices
  * Air-Q3 size 0 for neonates: < 2 kilograms
  * i-gel supraglottic airway size 1 for neonates: ≥ 2 kilograms
  Arms: Surfactant Administration through Laryngeal or Supraglottic Airway
Procedure: Surfactant Administration through Thin Catheter — Thin Catheter
  Arms: Surfactant Administration through Thin Catheter

SUMMARY:
What is this study about? This study is comparing two ways of giving surfactant, a medicine that helps premature infants breathe better. Surfactant can be given using a thin tube ("Less Invasive Surfactant Administration", called the LISA method) or through a small airway device placed in the baby's throat ("Surfactant Administration through Laryngeal or Supraglottic Airway", called the SALSA method). The goal is to see which method is safer and more effective for infants who are born at or after 29 weeks of pregnancy and have trouble breathing.

What is the main question (hypothesis)? Infants who receive surfactant using the SALSA method will have fewer breathing-related problems and fewer short-term complications than those who receive it using the LISA method.

What are the aims? Aim 1: Are babies in the SALSA group less likely to have low heart rate or low oxygen levels during the procedure compared to babies in the LISA group? Aim 2: Do fewer babies in the SALSA group need to be put on a breathing machine within the first 72 hours of life? Aim 3: Does the SALSA method help reduce the overall time babies need breathing support and lower the cost of their care in the NICU?

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants born at or greater than 29 weeks' gestational age
* Infants with birthweight greater than or equal to 750 grams and admitted to the NICU on CPAP for respiratory support and qualify for LISA procedure

Exclusion Criteria:

* Infants who require intubation prior to surfactant therapy
* Infants with known severe congenital anomalies (complex congenital heart disease, airway and central nervous system anomalies)
* Infants whose birth weight is less than 750 grams or oropharynx unable to accommodate laryngeal mask airways

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of events of bradycardia and hypoxemia during surfactant administration | Time of surfactant administration to completion of procedure
  * Bradycardia: defined as heart rate < 100 beats per minute for > 10 seconds. Heart rate will be obtained from participant's heart rate monitor.
  * Hypoxemia: oxygen saturation (SpO2) =< 80% for > 30 seconds. Oxygen saturation will be obtained from participant's pulse oximeter monitor
  * Events will be recorded by bedside respiratory therapy and/or bedside nurse during the procedure

SECONDARY OUTCOMES:
Procedural success rate on first attempt | At time of surfactant administration procedure
  * Procedure attempt is defined at the introduction of laryngoscope blade into mouth.
  * Procedural success is defined by the ability to insert catheter or laryngeal mask airway and administer surfactant without surfactant aspirated from the stomach post administration
  * Rate will be calculated as a percentage of participants in each arm
Intubation rate | From time of procedure to 72 hours of life
  * Rate will be calculated as a percentage of participants in each arm Invasive mechanical ventilation within first 72 hours of life after surfactant
  * Participants' need for and timing of intubation will be obtained from electronic medical record
Mean number of attempts required | At time of surfactant administration
  Procedure attempt will be defined as introduction of laryngoscope blade into mouth.
Total duration of CPAP and mechanical ventilation days | Up to 52 weeks
  Total numbers of days on continuous end positive expiratory pressure (CPAP) and invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Melody Chiu, M.D., Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No
Data will be collected and de-identified at the time of analysis. IPD availability does not to enhance study results.

REFERENCES:
- [Background] Roberts CT, Manley BJ, O'Shea JE, Stark M, Andersen C, Davis PG, Buckmaster A. Supraglottic airway devices for administration of surfactant to newborn infants with respiratory distress syndrome: a narrative review. Arch Dis Child Fetal Neonatal Ed. 2021 May;106(3):336-341. doi: 10.1136/archdischild-2020-319804. Epub 2020 Sep 28. PMID 32989046
- [Background] Roberts KD, Brown R, Lampland AL, Leone TA, Rudser KD, Finer NN, Rich WD, Merritt TA, Czynski AJ, Kessel JM, Tipnis SM, Stepka EC, Mammel MC. Laryngeal Mask Airway for Surfactant Administration in Neonates: A Randomized, Controlled Trial. J Pediatr. 2018 Feb;193:40-46.e1. doi: 10.1016/j.jpeds.2017.09.068. Epub 2017 Nov 22. PMID 29174079
- [Background] Wyckoff MH, Greif R, Morley PT, Ng KC, Olasveengen TM, Singletary EM, Soar J, Cheng A, Drennan IR, Liley HG, Scholefield BR, Smyth MA, Welsford M, Zideman DA, Acworth J, Aickin R, Andersen LW, Atkins D, Berry DC, Bhanji F, Bierens J, Borra V, Bottiger BW, Bradley RN, Bray JE, Breckwoldt J, Callaway CW, Carlson JN, Cassan P, Castren M, Chang WT, Charlton NP, Phil Chung S, Considine J, Costa-Nobre DT, Couper K, Couto TB, Dainty KN, Davis PG, de Almeida MF, de Caen AR, Deakin CD, Djarv T, Donnino MW, Douma MJ, Duff JP, Dunne CL, Eastwood K, El-Naggar W, Fabres JG, Fawke J, Finn J, Foglia EE, Folke F, Gilfoyle E, Goolsby CA, Granfeldt A, Guerguerian AM, Guinsburg R, Hirsch KG, Holmberg MJ, Hosono S, Hsieh MJ, Hsu CH, Ikeyama T, Isayama T, Johnson NJ, Kapadia VS, Kawakami MD, Kim HS, Kleinman M, Kloeck DA, Kudenchuk PJ, Lagina AT, Lauridsen KG, Lavonas EJ, Lee HC, Lin YJ, Lockey AS, Maconochie IK, Madar RJ, Malta Hansen C, Masterson S, Matsuyama T, McKinlay CJD, Meyran D, Morgan P, Morrison LJ, Nadkarni V, Nakwa FL, Nation KJ, Nehme Z, Nemeth M, Neumar RW, Nicholson T, Nikolaou N, Nishiyama C, Norii T, Nuthall GA, O'Neill BJ, Gene Ong YK, Orkin AM, Paiva EF, Parr MJ, Patocka C, Pellegrino JL, Perkins GD, Perlman JM, Rabi Y, Reis AG, Reynolds JC, Ristagno G, Rodriguez-Nunez A, Roehr CC, Rudiger M, Sakamoto T, Sandroni C, Sawyer TL, Schexnayder SM, Schmolzer GM, Schnaubelt S, Semeraro F, Skrifvars MB, Smith CM, Sugiura T, Tijssen JA, Trevisanuto D, Van de Voorde P, Wang TL, Weiner GM, Wyllie JP, Yang CW, Yeung J, Nolan JP, Berg KM; Collaborators. 2022 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations: Summary From the Basic Life Support; Advanced Life Support; Pediatric Life Support; Neonatal Life Support; Education, Implementation, and Teams; and First Aid Task Forces. Resuscitation. 2022 Dec;181:208-288. doi: 10.1016/j.resuscitation.2022.10.005. Epub 2022 Nov 3. PMID 36336195
- [Background] Kakkilaya V, Gautham KS. Should less invasive surfactant administration (LISA) become routine practice in US neonatal units? Pediatr Res. 2023 Apr;93(5):1188-1198. doi: 10.1038/s41390-022-02265-8. Epub 2022 Aug 19. PMID 35986148
- [Background] Kurepa D, Perveen S, Lipener Y, Kakkilaya V. The use of less invasive surfactant administration (LISA) in the United States with review of the literature. J Perinatol. 2019 Mar;39(3):426-432. doi: 10.1038/s41372-018-0302-9. Epub 2019 Jan 11. PMID 30635595
- [Background] Kakkilaya VB, Weydig HM, Smithhart WE, Renfro SD, Garcia KM, Brown CM, He H, Wagner SA, Metoyer GC, Brown LS, Kapadia VS, Savani RC, Jaleel MA. Decreasing Continuous Positive Airway Pressure Failure in Preterm Infants. Pediatrics. 2021 Oct;148(4):e2020014191. doi: 10.1542/peds.2020-014191. Epub 2021 Sep 22. PMID 34552000
- [Background] Committee on Fetus and Newborn; American Academy of Pediatrics. Respiratory support in preterm infants at birth. Pediatrics. 2014 Jan;133(1):171-4. doi: 10.1542/peds.2013-3442. Epub 2013 Dec 30. PMID 24379228